CLINICAL TRIAL: NCT04819464
Title: An Open-label, Parallel-group Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Cenerimod After Single-dose Administration in Subjects With Hepatic Impairment and in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics of a Single Dose of Cenerimod
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-064-106; 2020-006002-23 (EudraCT Number)
Record Dates: First submitted 2021-03-16; First posted 2021-03-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Hepatic Impairment
MeSH Terms: interventions — cenerimod

STUDY DESIGN:
Intervention Model Description: The 3 groups will be sequentially studied. Dosing will start in the participants with mild hepatic impairment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Participants with mild hepatic impairment (Experimental): Participants with mild hepatic impairment (Child-Pugh Score of 5 to 6).
  Interventions: Drug: Cenerimod
- Group B: Participants with moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh Score of 7 to 9).
  Interventions: Drug: Cenerimod
- Group C:Healthy participants (Experimental): Healthy participants will be matched to the participants with hepatic impairment based on age and body weight.
  Interventions: Drug: Cenerimod

INTERVENTIONS:
Drug: Cenerimod — A single oral dose of 0.5 mg.
  Other Names: ACT-334441

SUMMARY:
This is a prospective, open-label, single-dose, phase 1 study, to assess the effect of mild and moderate hepatic impairment on the pharmacokinetics of cenerimod (ACT-334441).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Women of child bearing potential must have a negative serum pregnancy test at screening, a negative urine pregnancy test on Day -1, and must agree to consistently and correctly use a highly effective method of contraception (i.e., failure rate of less than 1%).
* Women of non-childbearing potential must have a medical history of previous bilateral salpingectomy, salpingo-oophorectomy or hysterectomy, premature ovarian failure confirmed by a specialist gynecologist; or, be post-menopausal, defined as 12 consecutive months with amenorrhea prior to screening without alternative medical cause and confirmed with a follicle-stimulating hormone test.
* Body mass index of 18.0 to 32.0 kg/m2 (inclusive) at screening.
* Negative SARS-CoV-2-testing prior to Day -1 or documented vaccination against COVID-19 at least 3 months prior screening.
* Ability to communicate well with the investigator, in a language understandable to the participant, and to understand and comply with the requirements of the study.

Exclusion Criteria:

General (Group A, B and C)

* Pregnant or lactating women.
* Participation in a clinical study involving study treatment administration within 30 days prior to screening or in more than 2 clinical studies within 1 year prior to screening.
* Previous exposure to cenerimod.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, elimination (ADME) of the study treatment except for those related to liver cirrhosis or appendectomy and herniotomy.
* International Normalized Ratio greater than 2 at screening.
* Encephalopathy grade greater than or equal to 1.
* Clinically relevant abnormalities on a 12-lead ECG, recorded after 5 minutes in the supine position at screening and on Day 1 pre-dose.
* Presence of herpes simplex, disseminated zoster, or other opportunistic infections.
* Vaccination with live or live attenuated vaccines in the previous 4 weeks.
* Previous treatment with antiarrhythmic medications of class Ia or III 2 weeks or 5 half-lives, whichever is longer, prior to study treatment administration.
* Active retinopathy or macular edema at screening.
* Severe chronic obstructive pulmonary disease at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening.

Additional exclusion criteria for participants with hepatic impairment (Group A and B)

* Clinically relevant findings in clinical laboratory tests (hematology, coagulation, clinical chemistry, and urinalysis) at screening and on Day -1, except for those related to liver cirrhosis.

Additional exclusion criteria for healthy subjects (Group C)

* Clinically relevant findings in clinical laboratory tests (hematology, coagulation, clinical chemistry, and urinalysis) at screening and on Day -1.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St. John's Wort, homeopathic preparations, vitamins, and minerals) within 2 weeks or 5 t½ prior to study treatment administration, whichever is longer (excluding contraceptives and HRT).
* Aspartate aminotransferase and alanine aminotransferase above the upper limit of normal.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-08-18 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curves (AUC0-t): cenerimod | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Area under the plasma concentration-time curve from zero to infinity (AUC0-inf): cenerimod | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Maximum plasma concentration (Cmax): cenerimod. | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Time to reach Cmax (tmax): cenerimod | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Terminal half-life (t½): cenerimod | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Plasma protein binding of cenerimod | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Apparent clearance (CL/F) of cenerimod | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Apparent volume of distribution (Vz/F) of cenerimod | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 98.

SECONDARY OUTCOMES:
Total lymphocyte count | Multiple sampling at predefined times on Day 1 (pre-dose) up to Day 98.
Change from baseline at each time point of measurement in electrocardiogram QT interval | Pre-defined times on Day 1 (pre-dose) up to Day 105.
Change from baseline in body weight | Day -1 and Day 105.
Change from baseline in systolic and diastolic blood pressure (in the supine position) | Predefined times on Day 1 (pre-dose) up to Day 105.
Incidence of abnormal laboratory test results | Multiple sampling at predefined times on Day 1 (pre-dose) up to Day 105.
Adverse events and serious adverse events | Day 1 up to Day 105.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (2):
- CRU Hungary, Kistarcsa, Hungary
- BlueClinical Phase 1 Hospital de Prelado, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No